CLINICAL TRIAL: NCT01777048
Title: Augmenting the Effects of Methylphenidate: A Randomized, Placebo-Controlled Trial of Omega-3 Fatty Acids Supplementation in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Omega-3 Fatty Acids Supplementation in ADHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment numbers
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Universitäre Psychiatrische Kliniken (UPK) Basel (Unknown)
Responsible Party: Principal Investigator, Yoon Phaik Ooi, Researcher, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 203/12
Record Dates: First submitted 2013-01-16; First posted 2013-01-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 Fatty Acids (Experimental): 1g of Omega-3 per day [400mg DHA & 600mg EPA] for 12 weeks: 2 capsules after breakfast and 2 capsules after dinner
  Interventions: Dietary Supplement: Omega-3 Fatty Acids Supplementation
- Omega-3 Placebo (Placebo Comparator): 1g of Omega-3 Placebo per day for 12 weeks: 2 capsules after breakfast and 2 capsules after dinner
  Interventions: Dietary Supplement: Omega-3 Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids Supplementation
  Arms: Omega-3 Fatty Acids
Dietary Supplement: Omega-3 Placebo — Placebo capsules manufactured to mimic Omega-3 capsules
  Arms: Omega-3 Placebo

SUMMARY:
The overarching aim of the proposed study is to assess whether omega-3 fatty acids supplementation can augment the effects of methylphenidate in children with ADHD. The investigators hypothesized that omega-3 fatty acids supplementation will be associated with improved ADHD symptoms.

ELIGIBILITY:
Inclusion Criteria:

Participants between ages 6 and 12 years who:

1. have been clinically diagnosed with ADHD by a physician
2. meet the criteria of ADHD-Inattention, ADHD-Hyperactivity-Impulsivity, or ADHD-Combined type as determined by the SNAP-IV (Swanson, 1992)
3. are willing to participate in a randomized, double-blind, placebo-controlled trial, complete with written, informed parental consent,
4. are on stable dosage of methylphenidate treatment before the start of the study
5. are able to speak English or German

Exclusion Criteria:

1. Participants who are younger than 6 years old or older than 12 years old
2. Those who have not been clinically diagnosed with ADHD by a physician
3. Those who did not meet the criteria of ADHD-Inattention, ADHD-Hyperactivity-Impulsivity, or ADHD-Combined type as determined by the SNAP-IV (Swanson, 1992)
4. Those without written parental consent
5. Those with brain pathology such as serious head injury, epilepsy, and intellectual disability (IQ < 70)
6. Those with titrated dosage of methylphenidate before the start of the study
7. Those on neurofeedback training, and/or psychosocial intervention addressing attention problems
8. Those with known hypersensitivity to the IMP under investigation
9. Those who are unable to read and understand the parent/participant information
10. Those receiving medications other than methylphenidate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale-IV total score | Baseline, Week 6, and Week 12

SECONDARY OUTCOMES:
Change in Child Behaviour Checklist total score | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Phaik Ooi, PhD, Study Director — University of Basel
Locations (1):
- Universitäre Psychiatrische Kliniken (UPK) Basel, Basel, Switzerland

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600